CLINICAL TRIAL: NCT06097533
Title: Improvement of Quality of Life by Cannabinoids in Oncologic Patients (BEfindLichkeitsverbesserung Unter CANnabinoid-ExtrakTen Bei Onkologischen Patienten)
Brief Title: Improvement of Quality of Life by Cannabinoids in Oncologic Patients
Acronym: BELCANTO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Avextra Pharma GmbH (Unknown); SocraMetrics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BELCANTO; 2022-004137-39 (EudraCT Number); DRKS00031009 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Medical Oncology; Palliative Care; Quality of Life; Cannabinoids
Keywords: BELCANTO

STUDY DESIGN:
Intervention Model Description: Multi-center, prospective, interventional, randomized, two-arm, placebo-controlled, parallel, double-blinded clinical trial according to German Drug Law (AMG)/GCP and German Narcotic Drugs Act (BtMG)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: IMPs are centrally blinded and randomised at the pharmacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabisextrakt Avextra 10/10 Lösung (Experimental): Solution with tetrahydrocannabinol and cannabidiol
  Interventions: Drug: Cannabisextrakt Avextra 10/10 Lösung
- Placebo (Placebo Comparator): Sesame oil, Ph.Eur. Linseed oil, Ph.Eur
  Interventions: Drug: Cannabisextrakt Avextra 10/10 Lösung

INTERVENTIONS:
Drug: Cannabisextrakt Avextra 10/10 Lösung — medical cannabinoids
  Other Names: Cannabisextrakt Avextra 10/10 solution

SUMMARY:
The goal is to explore whether the application of cannabis extract Avextra 10/10 solution is suitable to contribute to an improvement in the symptom burden and well-being of oncological palliative care patients. The primary objective of the study is to demonstrate the improvement in global symptom burden in the intervention arm compared to the placebo control group over a period of 12±2 days, as measured by a percentage change in the value of the Edmonton Symptom Assessment System total symptom distress score (ESAS TSDS) at baseline and after 12±2 days.

DETAILED DESCRIPTION:
170 oncological patients in palliative treatment will be randomized 1:1 to an THC:CBD-interventional arm and an placebo-arm. At the timepoints baseline, 12±2 days, 18±3 days, four weeks and eight weeks, the global burden of symptoms (ESAS TSDS), quality of life (EORTC QLQ C15 PAL) and other parameter will be measured and the intraindividual difference in comparison with the baseline will be compared between the groups. This study is intended to provide a significant contribution to Evidence-based medicine (EbM) of CAM in palliative medicine as well as for elderly and severely ill subjects (resp.) in general.

The following gain of knowledge is expected:

* substancial and reliable effects of CAM in elderly subjects being in a multimorbid and psychologically very stressful situation of illness and life (resp.).
* substancial and reliable effects of CAM in aduld subjects being in a oncologically and palliative situation of illness and life (resp.).
* compatibility of a CAM-therapy in multimorbid patients with polypharmacotherapy.
* importance of CAM for the very frequent psychovegetative disturbance and comorbidities of many illnesses like sleepnesness, loss of appetite, nausea, fear and affective disturbance.
* possible reduction of costs and improved economics through CAM

ELIGIBILITY:
Inclusion Criteria:

* ≥25 years old and legally competent
* Palliative oncological therapy
* ECOG status 1, 2 or 3, incapacitated for work
* ESAS TSDS > or equals 16
* Nutritional Risk Screening > or equals 3
* Pain numerical rating scale > or equals 4
* informed consent
* for WOCBP:

  * Negative pregnancy test
  * Reliable contraception (Pearl Index < 1%)

Exclusion Criteria:

* nausea > or equals grade 3 (CTCAE) or vomiting > or equals grade 2 (CTCAE) in the preceding week
* Inability to understand and complete the questionnaires
* Cannabis use in the last 6 weeks
* Alcohol addiction
* Pregnancy/lactation
* Contraindications or intolerance to the study medication (esp. psychosis)
* Simultaneous participation in other clinical studies (sumulataneous participation in non-interventional studies (i.e. biomarker-studies, registries) is allowed, if the study-aim does not interfere with measures of the second study)
* Any other condition as judged by the investigator, e.g. non-compliance

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
ESAS-TSDS score | 12 days
  Symptom change as percentage change in ESAS-TSDS score after 12±2 days compared to baseline between intervention group and placebo control group.

SECONDARY OUTCOMES:
Global Patient's Assessment | 12 days, 4 weeks, 8 weeks
  Scale to evaluate the absolute severity and the change in comparison with the preceding measurement
opioid dose as morphine equivalent | 12 days, 4 weeks, 8 weeks
defined daily dosages (DDD) of neuropharmaceuticals | 12 days, 4 weeks, 8 weeks
ESAS-TSDS score | 4 weeks, 8 weeks
  Edmonton Symptom Assessment System
inappetence | 12 days, 4 weeks, 8 weeks
NCCN distress thermometer | 12 days, 4 weeks, 8 weeks
pain as VAS | 12 days, 4 weeks, 8 weeks
sleep quality (Pittsburgh Sleep Quality Index, PSQI) | 12 days, 4 weeks, 8 weeks
  contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available)
EORTC QLQ-C15 PAL | 12 days, 4 weeks, 8 weeks
  European Organization for Research and Treatment of Cancer Quality of Life Palliative
Adverse events (AE) | up to 8 weeks
  Adverse events (AE) incidence, frequency and severity coded according to the Medical Dictionary for Regulatory Activities (MedDRA) and scored according to the NCI Common Terminology Criteria for Adverse Events (CTCAE)
C-reactive protein (CRP) | 12 days, 4 weeks, 8 weeks
all endpoints stratified by stage of oncological disease (ICD-10), treatment modalities, gender, weight, high/low dose, renal function and age whereever possible and meaningful | 12 days, 4 weeks, 8 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Hubertus Wald Tumorzentrum Universitäres Cancer Center Hamburg (UCCH), Hamburg, Hamburg
  - University Hospital Schleswig-Holstein, Kiel, Schleswig-Holstein
  - University Hospital Schleswig-Holstein, Lübeck, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: Undecided
Aggregated data can be shared. Individual data only after internal and IRB review.